CLINICAL TRIAL: NCT03977077
Title: A Retrospective Clinical Study on the Efficacy and Safety of Injection Taxol (Albumin Binding Type) in the Treatment of Patients With Advanced Gastrointestinal Tumors
Brief Title: Treatment of Advanced Gastrointestinal Tumors With Albumin Taxol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AYGAS-0531
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-05

CONDITIONS: Advanced Gastrointestinal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albumin binding taxol (Experimental)
  Interventions: Drug: Albumin binding taxol

INTERVENTIONS:
Drug: Albumin binding taxol — 125mg/m2, d1, 8, intravenous infusion for 30min, 1 cycle every 3 weeks;Other combined chemotherapy drugs and drug doses shall be administered by clinicians according to the guidelines and the actual situation of clinical patients.

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of domestic injection paclitaxel (albumin binding type) in patients with advanced digestive tract tumors,and to further explore the possible predictors of efficacy.In order to provide more effective chemotherapeutic drugs, prolong survival time and improve quality of life for patients with advanced digestive tract tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years with advanced esophageal cancer, gastric cancer, pancreatic cancer and gallbladder (duct) confirmed histologically by albumin paclitaxel chemotherapy regimen;
2. ECOG PS 0-2；
3. Expected survival time ≥3 months;
4. According to RECIST1.1, at least one measurable lesion exists；
5. The level of organ function must meet the following requirements（1）Blood routine examination standards must be met：HB≥90 g/L；ANC≥1.5×109/L； PLT≥80×109/L；（2）Liver function should meet the following criteria TBIL≤1.5×ULN；AST≤2.5×ULN；（3）Renal function should meet the following criteria: CrCL≥60 ml/min；

Exclusion Criteria:

1. Pregnant or lactating women；
2. Had a history of other primary malignancies within 5 years, with the exception of cured basal cell skin cancer and cured cervical cancer;
3. Active brain metastasis or severe disease;
4. Grade 1 peripheral neuropathy (judged according to NCICTC standard for adverse reactions);
5. Patients with allergy to research drugs, albumin or previous allergies;
6. Severe mental or neurological disorders affecting the presentation or observation of adverse reactions;
7. The investigator considers that there is any condition that may impair the subject or cause the subject to fail to meet or perform the study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to 2 year
  Progression free survival (PFS) is the time between the onset of treatment and the observation of disease progression or death from any cause.

SECONDARY OUTCOMES:
Objective remission rate (ORR) | up to 2 year
  Defined as the proportion of patients with a documented complete response, and partial response (CR+PR)
Overall survival | up to 2 year
  The Overall survival (OS) is defined as the date from random grouping to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China